CLINICAL TRIAL: NCT03182790
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2017: a Single-blind Cluster Randomized Controlled Trial on a Combined "Cocktail" Intervention of Brief Advice, Instant Messaging and Active Referral (AIR) to Increase Abstinence
Brief Title: Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW 2017
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Quit to Win; Brief intervention; Semi-personalized Instant messaging; Incentives; AWARD model; Smoking Cessation Intervention; Regular messages
MeSH Terms: conditions — Smoking Cessation | interventions — corticosteroid hormone-induced factor; Referral and Consultation; Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Instant Messaging IM + regular messages +AWARD advice + warning leaflet + referral card
  Interventions: Behavioral: Instant Messaging IM; Behavioral: Regular messages; Behavioral: AWARD advice; Behavioral: Referral card; Behavioral: COSH booklet; Behavioral: Warning Leaflet
- Group B (Experimental): COSH booklet + general brief advices +Placebo Messages
  Interventions: Behavioral: Brief advice; Behavioral: COSH booklet; Behavioral: Placebo Messages

INTERVENTIONS:
Behavioral: Instant Messaging IM — Smokers can communicate with counsellors in real-time through instant messaging (social media). Our counsellors will trigger the conversation and invite the smokers to response after initial contact. Counsellors will keep contact with the smokers to offer help, positive encouragement, reflections and reminders about SC according to smokers' personal needs and to encourage them to seek SC services. Details of successfully booked SC appointment (e.g. SC services address, contact information, date, appointment number etc.) will be delivered to the smokers using IM. All smokers will receive a reminder-to-attend IM messages 1-3 days before the appointment date.
  Other Names: Instant messaging interaction
  Arms: Group A
Behavioral: Regular messages — Regular messages, including: harm of smoking, benefit of smoking cessation, importance of adherence to smoking cessation appointment and encouragement on abstinence will be sent to smokers after initial contact via social media.
  Other Names: Regular messages focusing active referral and encouragement
  Arms: Group A
Behavioral: AWARD advice — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again (if the smokers refused to set quit date).
  Other Names: Ask, Warn, Advise, Refer, Do-it-again
  Arms: Group A
Behavioral: Referral card — The 3-folded "Smoking Cessation Services" card consists of brief information and highlights of existing smoking cessation services, contact methods, motivation information and strong supporting messages or slogans
  Other Names: Smoking Cessation Service Card
  Arms: Group A
Behavioral: Brief advice — Very brief, minimal and general smoking cessation advice
  Other Names: Brief smoking cessation advice
  Arms: Group B
Behavioral: COSH booklet — A general smoking cessation self-help booklet
  Other Names: COSH self-help smoking cessation booklet
Behavioral: Placebo Messages — Placebo messages will be sent via smart phones (e.g. social media) to remind subjects to take follow-up calls before each follow-up time points.
  Arms: Group B
Behavioral: Warning Leaflet — The leaflet will include the information about the health risks of smoking.
  Arms: Group A

SUMMARY:
The present study will examine (1) the effectiveness of regular messages and semi-personalized instant messaging with AWARD brief advice and active referral to smoking cessation (SC) services and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

DETAILED DESCRIPTION:
Although smoking prevalence is decreasing in Hong Kong, there are still 641,300 daily smokers (10.5%) and half will be killed by smoking which accounts for over 7,000 deaths per year. Smoking also accounts for a large amount of medical cost, long-term care and productivity loss of US$688 million (0.6% Hong Kong GDP). Smoking is a highly addictive behavior and it is difficult for smokers with strong nicotine dependence to quit without assistance. On the other hand, reaching and helping the many smokers who have no intention to quit is a challenge, because they are unlikely to seek professional help from smoking cessation services.

The Quit and Win programme provides an opportunity to reach and encourage a large group of smokers to make quit attempt and maintain abstinence. The Quit and Win model posits that smokers participating in the contest will have higher motivation to quit with incentives and better social support. Studies have found that such quitting contests or incentive programs appeared to reach a large number of smokers and demonstrated a significantly higher quit rate for the quit and win group than for the control group.

Smoking cessation services in Hong Kong are under-used with most of the adult daily smokers (79.6%) who had never used smoking cessation services. Among these smokers, only 2.4% were willing to use the services. Our previous RCT in previous QTW Contest 2015 evaluated the effects of low-intensity active referral (LAR) vs. very brief general SC advice (VBA) on quitting. LAR included onsite AWARD counselling and collection of smokers' personal contact information for SC services providers to connect with the smokers. Findings at 3-month follow-up of this RCT suggested the LAR intervention resulted in significantly higher self-reported quit rate than VBA in the control group (18.7% vs. 14.0%. P<0.001). Our RCT in previous QTW Contest 2016 evaluated the effects of a higher intensity and personalized active referral (HAR) vs. low intensity text messaging (SMS) vs. very brief SC advice (VBA; control group) on encouraging smoking cessation (SC) service use and increasing the quit rate. Findings at 6-month follow-up of the QTW 2016 RCT showed that the intervention group with HAR had a significantly higher self-reported quit rate than VBA (the control group) (17.0% vs. 11.2%, P = 0.02). Text messaging group also had significantly higher self-reported quit rate than the control group (17.1 % vs. 11.2%, P = 0.02).

However, these SMS-based RCTs could not provide real-time responses from the counsellors, which might weaken the smokers' intention to quit and lower the intensity of social support. In the present proposal, we hope to enrich the SMS-based intervention by using social media such as WhatsApp or WeChat etc., which can provide an interactive platform and develop a semi-personalized interactive IM system that can tailor for the smokers according to their characteristics, needs and demand.

Therefore, the present study will examine (1) the effectiveness of regular messages and semi-personalized instant messaging with AWARD brief advice and active referral to smoking cessation (SC) services and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese (including reading Chinese)
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO Smokerlyzer.
* Intent to quit / reduce smoking
* Using a cell phone with instant messaging tool (e.g. WhatsApp, WeChat)
* Able to use instant messaging tool (e.g. WhatsApp, WeChat) for communication

Exclusion Criteria:

* Smokers who have communication barrier (either physically or cognitively)
* Have participation in other smoking cessation programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1311 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Biochemical validated quit rate at 6-month follow-up | 6-month follow-up
  Biochemically validated quit rates at 6-month in the two groups

SECONDARY OUTCOMES:
Biochemical validated quit rate | 3-month follow-up
  Biochemically validated quit rates at 3-month in the two groups
Smoking quit rate change from baseline at 3-month follow-up | 3-month follow-up
  The primary outcomes are self-reported 7-day point prevalence (pp) quit rate at 3-month between the two groups
Smoking quit rate change from baseline at 6-month follow-up | 6-month follow-up
  The primary outcomes are self-reported 7-day point prevalence (pp) quit rate at 6-month between the two groups
Smoking reduction rate change from baseline at 3-month follow-up | 3-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Smoking reduction rate change from baseline at 6-month follow-up | 6-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Smoking quit attempt change from baseline at 3-month follow-up | 3-month follow-up
  Number of quit attempts at 3-month in the two groups
Smoking quit attempt change from baseline at 6-month follow-up | 6-month follow-up
  Number of quit attempts at 6-month in the two groups
Quit rate for all subjects change from baseline at 3- and 6-month follow-up | 3 and 6 months follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2017
Reduction rate for all subjects change from baseline at 3- and 6-month follow-up | 3 and 6 months follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2017
Use of smoking cessation service | 3 and 6 months follow-up
  Use of smoking cessation at 3 and 6 month follow-up in the two groups
Use of smoking cessation service for all subjects | 3 and 6 months follow-up
  Use of smoking cessation service for all subjects participating in Quit to Win contest 2017

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Kelvin Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Council on Smoking and Health (COSH), Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Luk TT, Cheung YTD, Zhao S, Zeng Y, Tong HSC, Lai VWY, Wang MP. Engagement With a Mobile Chat-Based Intervention for Smoking Cessation: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2417796. doi: 10.1001/jamanetworkopen.2024.17796. PMID 38922618
- [Derived] Wang MP, Luk TT, Wu Y, Li WH, Cheung DY, Kwong AC, Lai V, Chan SS, Lam TH. Chat-based instant messaging support integrated with brief interventions for smoking cessation: a community-based, pragmatic, cluster-randomised controlled trial. Lancet Digit Health. 2019 Aug;1(4):e183-e192. doi: 10.1016/S2589-7500(19)30082-2. Epub 2019 Jul 31. PMID 33323188